CLINICAL TRIAL: NCT02532244
Title: Genetics of Pediatric-Onset Motor Neuron and Neuromuscular Diseases
Status: Completed | Type: Observational
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Matthew E. R. Butchbach, Ph.D., Research Scientist, Nemours Children's Clinic
Other Study IDs: 764456
Record Dates: First submitted 2015-08-21; First posted 2015-08-25 (Estimated); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Spinal Muscular Atrophy; Charcot-Marie-Tooth Disease; Muscular Dystrophy; Spinal Muscular Atrophy With Respiratory Distress 1; Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Neuromuscular Disease; Peroneal Muscular Atrophy
Keywords: distal hereditary motor neuronopathy
MeSH Terms: conditions — Muscular Atrophy, Spinal; Charcot-Marie-Tooth Disease; Muscular Dystrophies; Spinal muscular atrophy with respiratory distress 1; Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Neuromuscular Diseases | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, lymphoblastoid cell lines derived from peripheral blood mononuclear cells, saliva, buccal cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sample collection: Each participant will have blood drawn for genetic analysis and for establishment of a lymphoblastoid cell line.
  Interventions: Other: sample collection

INTERVENTIONS:
Other: sample collection — collection of blood

SUMMARY:
The goal of this study is to establish a genetic registry of patients with early-onset motor neuron and neuromuscular diseases. The investigators will collect samples from patients with a motor neuron or a neuromuscular disorder and their family members. The samples to be collected will be obtained using minimally invasive (whole blood) means. The research team will then extract high quality genomic DNA or RNA from these samples and use it to identify and confirm novel gene mutations and to identify genes which regulate the severity of motor neuron/neuromuscular diseases.

DETAILED DESCRIPTION:
Diseases affecting the motor unit--which is composed of the motor neuron, its myelin sheath and its innervated muscle fibers--are a diverse, heterogeneous group having heterogeneous clinical presentations and genetic causes. Many of these disorders have a inherited component. In some cases, the genetics underlying a given neuromuscular/motor neuron disease, like spinal muscular atrophy (SMA) or Duchenne muscular dystrophy, are well characterized. There are, however, disorders whose genetic basis has yet to be determined or genetically characterized diseases which harbor novel mutations. The purpose of this genetic registry is to catalogue early-onset motor neuron and neuromuscular disorders and to determine their genetic bases. With samples obtained from this registry, the investigators will be able to provide a genetic diagnosis for a specific neuromuscular/motor neuron disease which will lead to better care for those patients affected by these diseases.

Many of these disorders have a wide spectrum of phenotypic variability. For example, the severity of SMA is quite variable even though it is caused by the loss of a single gene, i.e. survival motor neuron 1 (SMN1). The number of copies of the duplicated gene survival motor neuron 2 (SMN2) dictates phenotypic severity in SMA. In this study, the research team will also identify potential modifiers of phenotypic severity for specific disorders like SMA and Charcot-Marie-Tooth (CMT) disease. With the identification of novel modifier genes, the investigators will be able to more accurately predict disease outcomes and the investigators will also have novel targets for the development of therapeutic agents for these diseases.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of motor neuron/neuromuscular disease confirmed by neurologist
* Be seen by one of the study investigators

Exclusion Criteria:

* not seen by one of the study investigators

Min Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will enroll children diagnosed with a motor neuron or neuromuscular disease as well as their parents and/or siblings as well as adults with childhood-onset motor neuron or neuromuscular diseases.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
genetic diagnosis | up to 2 years
  The genetic basis for the subject's condition will be verified/determined by Sanger sequencing of DNA sample

SECONDARY OUTCOMES:
SMN1 copy number | up to 2 years
  The number of copies of the SMN1 gene will be determined using array digital polymerase chain reaction (PCR).
SMN2 copy number | up to 2 years
  The number of copies of the SMN2 gene will be determined using array digital PCR.
target gene mRNA levels | up to 2 years
  The relative levels of the disease gene-specific messenger ribonucleic acid (mRNA) will be measured using quantitative PCR.
target gene protein levels | up to 2 years
  The relative amounts of the disease-gene-specific protein will be measured using immunoblot.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew ER Butchbach, Ph.D., Principal Investigator — Nemours Children's Clinic
Locations (3):
- United States (3):
  - Nemours Children's Hospital Delaware, Wilmington, Delaware
  - Nemours Children's Specialty Care, Jacksonville, Florida
  - Nemours Children's Hospital Orlando, Orlando, Florida

IPD SHARING:
Plan to Share IPD: Undecided
De-identified information will be shared once the data are published.

REFERENCES:
- [Result] Stabley DL, Holbrook J, Harris AW, Swoboda KJ, Crawford TO, Sol-Church K, Butchbach MER. Establishing a reference dataset for the authentication of spinal muscular atrophy cell lines using STR profiling and digital PCR. Neuromuscul Disord. 2017 May;27(5):439-446. doi: 10.1016/j.nmd.2017.02.002. Epub 2017 Feb 6. PMID 28284873
- [Result] Stabley DL, Harris AW, Holbrook J, Chubbs NJ, Lozo KW, Crawford TO, Swoboda KJ, Funanage VL, Wang W, Mackenzie W, Scavina M, Sol-Church K, Butchbach ME. SMN1 and SMN2 copy numbers in cell lines derived from patients with spinal muscular atrophy as measured by array digital PCR. Mol Genet Genomic Med. 2015 Jul;3(4):248-57. doi: 10.1002/mgg3.141. Epub 2015 Mar 21. PMID 26247043
- [Result] Chen X, Sanchis-Juan A, French CE, Connell AJ, Delon I, Kingsbury Z, Chawla A, Halpern AL, Taft RJ; NIHR BioResource; Bentley DR, Butchbach MER, Raymond FL, Eberle MA. Spinal muscular atrophy diagnosis and carrier screening from genome sequencing data. Genet Med. 2020 May;22(5):945-953. doi: 10.1038/s41436-020-0754-0. Epub 2020 Feb 18. PMID 32066871
- [Result] Jiang L, Lin R, Gallagher S, Zayac A, Butchbach MER, Hung P. Development and validation of a 4-color multiplexing spinal muscular atrophy (SMA) genotyping assay on a novel integrated digital PCR instrument. Sci Rep. 2020 Nov 16;10(1):19892. doi: 10.1038/s41598-020-76893-7. PMID 33199817
- [Result] Stabley DL, Holbrook J, Scavina M, Crawford TO, Swoboda KJ, Robbins KM, Butchbach MER. Detection of SMN1 to SMN2 gene conversion events and partial SMN1 gene deletions using array digital PCR. Neurogenetics. 2021 Mar;22(1):53-64. doi: 10.1007/s10048-020-00630-5. Epub 2021 Jan 7. PMID 33415588
- [Result] Pinto A, Cunha C, Chaves R, Butchbach MER, Adega F. Comprehensive In Silico Analysis of Retrotransposon Insertions within the Survival Motor Neuron Genes Involved in Spinal Muscular Atrophy. Biology (Basel). 2022 May 27;11(6):824. doi: 10.3390/biology11060824. PMID 35741345